CLINICAL TRIAL: NCT02223117
Title: Evaluation of the Safety and Immunogenicity of Autologous Thrombosomes® in Healthy Human Subjects; A Microdose Escalation Study (Cohorts 1 - 4) and Repeat Microdose Immunogenicity Study (Cohort 5)
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Cellphire Therapeutics, Inc. (Industry)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2011-1
Record Dates: First submitted 2014-08-15; First posted 2014-08-22 (Estimated); Last update posted 2017-12-13 (Actual); Status verified 2017-12

CONDITIONS: Healthy
MeSH Terms: interventions — Buffers

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Thrombosomes
  Interventions: Biological: Thrombosomes
- Placebo (Placebo Comparator): Buffer/placebo Control
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Thrombosomes — Freeze-dried platelets
  Arms: Intervention
Biological: Placebo
  Other Names: Buffer/placebo Control
  Arms: Placebo

SUMMARY:
This "first-in-human" exploratory IND, single-center study will assess the safety, toxicity, hematology, and immunogenicity of sub-therapeutic "microdoses" of autologous Thrombosomes® in healthy human subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Minimum weight 110 pounds (50 kg)
2. Age 18-45 years
3. Able and willing to provide informed consent
4. Has permanent address and phone/e-mail for contact and notification, and able to come to the research site for scheduled study visits for up to 60 days after their last study infusion
5. Understands, speaks and reads standard English language
6. Normal healthy subject able to pass the universal blood donor history questionnaire and screen

Exclusion Criteria:

1. Breast-feeding female
2. At any time, previously pregnant female
3. Participation in an experimental drug/device study within the past 30 days.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2016-07-21 (Actual); Study Completion 2016-07-21 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety Evaluation | 60 days

SECONDARY OUTCOMES:
Standard Hematology, Coagulation and Platelet Immunology Assessment | 60 Days

CONTACTS AND LOCATIONS:
Overall Officials: Michael Fitzpatrick, PhD, Study Director — Cellphire Therapeutics, Inc.; Sherrill Slichter, MD, Principal Investigator — Bloodworks Northwest
Locations (1):
- Bloodworks Northwest, Seattle, Washington, United States